CLINICAL TRIAL: NCT04148300
Title: The Impact of Oral Health Literacy on Dental Anxiety and Utilization of Oral Health Services Among Dental Patients: A Cross Sectional Study
Brief Title: The Impact of Oral Health Literacy on Dental Anxiety and Utilization of Oral Health Services
Status: Completed | Type: Observational
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Other Study IDs: PUB2121002
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2020-10

CONDITIONS: Oral Health
Keywords: Oral health literacy; Dental anxiety; Utilization of oral health services; Dental patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Oral Health Literacy is an integral part that should be taken into measures when evaluating the oral health status of any population. It has been stated that adults with low oral health literacy are more prone to miss their dental appointments and that low levels of oral health literacy, and being anxious and fearful of the dentist is a common barrier to the utilization of dental services. Unfortunately no previous studies assessed the oral health literacy level, dental anxiety and utilization of dental services among the Egyptian population. So the aim of the current study is to detect the impact of oral health literacy on level of dental anxiety and utilization of dental services among Misr International University (MIU) dental patients.

DETAILED DESCRIPTION:
The current study is a cross sectional study that includes an interview lead questionnaire that will be carried out by second year dental students of the academic years (2018-2019, 2019- 2020). The questionnaire consists of four sections; a demographic section, a modified Arabic Rapid Estimate of Adult Literacy (ARELAD-30) Tool, Arabic Modified Dental Anxiety Scale (AMDAS), and Utilization of oral health services questionnaire. Before conducting the study, orientation sessions and thorough training of the students will be performed to ensure that the students can conduct the interview consistently and efficiently. Students will be asked to design educational materials (brochures, leaflets and posters) that aim at improving patients' knowledge and awareness regarding oral health and the utilization of oral health services. The aim of this study is to detect the impact of oral health literacy on the level of dental anxiety and utilization of dental services among dental patients.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age: 18 - 60 years old.
* Dentate or partially edentulous patients with or without fixed or removable appliances.
* Healthy adults as well as adults with any chronic condition and/or under regular use of medication.

Exclusion Criteria:

* Subjects with mental or psychological problems.
* Subjects who cannot read or write.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Dental patients of both gender, aged from 18-60 years old, who can read.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Level of Oral Health Literacy | 14 months from the first enrollment
  modified version of the Arabic Version of Rapid Estimate of Adult Literacy in Medicine (AREALD-30): grades 0 (Complete illiteracy)-30 (Complete literacy)

SECONDARY OUTCOMES:
Level of Dental Anxiety | 14 months from the first enrollment
  Arabic Modified Dental Anxiety Scale (AMDAS): Likert scale 1(Extreme anxiety) -5 (Not anxious at all)
Level of utilization of oral health services | 14 months from the first enrollment
  Questionnaire: Nominal outcome (%)

CONTACTS AND LOCATIONS:
Overall Officials: Mahassen M. Farghaly, Professor, Study Director — Vice President for Community Services & Environmental Affairs
Locations (1):
- Faculty of Oral & Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo Y, Logan HL, Dodd VJ, Muller KE, Marks JG, Riley JL 3rd. Health literacy: a pathway to better oral health. Am J Public Health. 2014 Jul;104(7):e85-91. doi: 10.2105/AJPH.2014.301930. Epub 2014 May 15. PMID 24832423
- [Background] Batista MJ, Lawrence HP, Sousa MDLR. Oral health literacy and oral health outcomes in an adult population in Brazil. BMC Public Health. 2017 Jul 26;18(1):60. doi: 10.1186/s12889-017-4443-0. PMID 28747157
- [Background] Bahammam MA, Hassan MH. Validity and reliability of an Arabic version of the modified dental anxiety scale in Saudi adults. Saudi Med J. 2014 Nov;35(11):1384-9. PMID 25399217
- [Background] Saatchi M, Abtahi M, Mohammadi G, Mirdamadi M, Binandeh ES. The prevalence of dental anxiety and fear in patients referred to Isfahan Dental School, Iran. Dent Res J (Isfahan). 2015 May-Jun;12(3):248-53. PMID 26005465
- [Background] Fayad MI, Elbieh A, Baig MN, Alruwaili SA. Prevalence of Dental Anxiety among Dental Patients in Saudi Arabia. J Int Soc Prev Community Dent. 2017 Mar-Apr;7(2):100-104. doi: 10.4103/jispcd.JISPCD_19_17. Epub 2017 Mar 29. PMID 28462178
- [Background] Tadakamadla SK, Quadri MF, Pakpour AH, Zailai AM, Sayed ME, Mashyakhy M, Inamdar AS, Tadakamadla J. Reliability and validity of Arabic Rapid Estimate of Adult Literacy in Dentistry (AREALD-30) in Saudi Arabia. BMC Oral Health. 2014 Sep 29;14:120. doi: 10.1186/1472-6831-14-120. PMID 25267119
- [Background] Bommireddy VS, Koka KM, Pachava S, Sanikommu S, Ravoori S, Chandu VC. Dental Service Utilization: Patterns and Barriers among Rural Elderly in Guntur District, Andhra Pradesh. J Clin Diagn Res. 2016 Mar;10(3):ZC43-7. doi: 10.7860/JCDR/2016/17834.7456. Epub 2016 Mar 1. PMID 27135000
- [Background] Crego A, Carrillo-Diaz M, Armfield JM, Romero M. From public mental health to community oral health: the impact of dental anxiety and fear on dental status. Front Public Health. 2014 Feb 28;2:16. doi: 10.3389/fpubh.2014.00016. eCollection 2014. PMID 24616889
- [Background] Burgette JM, Lee JY, Baker AD, Vann WF Jr. Is Dental Utilization Associated with Oral Health Literacy? J Dent Res. 2016 Feb;95(2):160-6. doi: 10.1177/0022034515617457. Epub 2015 Nov 13. PMID 26567035